CLINICAL TRIAL: NCT03082586
Title: Phase I Trial of Radiation Dose Escalation With Concurrent Weekly Cisplatin and Paclitaxel in Patients With Esophageal Cancer
Brief Title: Radiation Dose Escalation in Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chen tingfeng, Director,department of radiation, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGH201705
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-06

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- radiochemotherapy 1 (Experimental): Patients will be treated with radiation therapy 57.2 Gy.
  Interventions: Radiation: radiochemotherapy 1
- radiochemotherapy 2 (Experimental): Patients will be treated with radiation therapy 64.4 Gy.
  Interventions: Radiation: radiochemotherapy 2
- radiochemotherapy 3 (Experimental): Patients will be treated with radiation therapy 71.6 Gy.
  Interventions: Radiation: radiochemotherapy 3
- radiochemotherapy 4 (Experimental): Patients will be treated with radiation therapy 78.8 Gy.
  Interventions: Radiation: radiochemotherapy 4
- radiochemotherapy 5 (Experimental): Patients will be treated with radiation therapy 86 Gy.
  Interventions: Radiation: radiochemotherapy 5
- radiochemotherapy 6 (Experimental): Patients will be treated with radiation therapy 93.2 Gy.
  Interventions: Radiation: radiochemotherapy 6

INTERVENTIONS:
Radiation: radiochemotherapy 1 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 7.2 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2, weekly; paclitaxel, 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen
  Arms: radiochemotherapy 1
Radiation: radiochemotherapy 2 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 14.4 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen
  Arms: radiochemotherapy 2
Radiation: radiochemotherapy 3 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 21.6 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen
  Arms: radiochemotherapy 3
Radiation: radiochemotherapy 4 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 28.8 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen
  Arms: radiochemotherapy 4
Radiation: radiochemotherapy 5 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 36 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
  Other Names: concurrent chemoradiotherapy regimen
  Arms: radiochemotherapy 5
Radiation: radiochemotherapy 6 — concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 43.2 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
  Other Names: concurrent chemoradiotherapy regimen
  Arms: radiochemotherapy 6

SUMMARY:
The aim of this trial is to find the maximum tolerable dose of radiation that can be delivered combined with chemotherapy (DDP & Paclitaxel) in patients with inoperable or medically unresectable esophageal cancer.

DETAILED DESCRIPTION:
The RTOG 8501 has established concurrent radiochemotherapy as the standard of care for cancer of the esophagus.However, locoregional remain problematic, with 25% of patients having persistence and 20% relapse of locoregional disease following the combined modality approach. New regimen is urgently needed for improving localregional control and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary squamous cell carcinoma of the esophagus
2. Age 1 8-75.
3. Patients must be deemed unresectable disease or patient is not deemed operable due to medical reasons.
4. Patients with distant metastasis and life expectancy >/= 3 months are eligible.
5. Zubrod performance status 0 to 2
6. No prior radiation to the thorax that would overlap with the current treatment field.
7. Patients with nodal involvement are eligible
8. Adequate bone marrow, renal and hepatic functions as assessed by the following: Hemoglobin >/= 10.0 g/dl, Platelet count >/= 1 00,000/mm^3,absolute granulocyte count (AGC) ≥2 × 10^9 cells/L,bilirubin and Aspartate transaminase ≤1.5 ×upper limit of normal (ULN), Creatinine </=1 .5 times ULN.
9. A signed informed consent must be obtained prior to therapy. 1 0. Induction chemotherapy is allowed.

Exclusion Criteria:

1. The presence of a fistula.
2. Prior radiotherapy that would overlap the radiation fields.
3. gastroesophageal junction cancer.
4. Uncontrolled concurrent illness including, but not limited to: Chronic Obstructive Pulmonary Disease(COPD) exacerbation or other respiratory illness, serious uncontrolled infection, symptomatic congestive heart failure (CHF),unstable angina pectoris, uncontrolled hypertension,or psychiatric illness/social situations that would limit compliance with the study requirements.
5. Known hypersensitivity to paclitaxel.
6. Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.
7. Acquired Immune Deficiency Syndrome.
8. Conditions precluding medical follow-up and protocol compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tingfeng Chen, MD, Principal Investigator — the ethic committee of shanghai genernal hospital
Locations (1):
- the Ethic Committee of Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Background] Herskovic A, Martz K, al-Sarraf M, Leichman L, Brindle J, Vaitkevicius V, Cooper J, Byhardt R, Davis L, Emami B. Combined chemotherapy and radiotherapy compared with radiotherapy alone in patients with cancer of the esophagus. N Engl J Med. 1992 Jun 11;326(24):1593-8. doi: 10.1056/NEJM199206113262403. PMID 1584260

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiochemotherapy 1 | Radiochemotherapy 2 | Radiochemotherapy 3 | Radiochemotherapy 4 | Radiochemotherapy 5 | Radiochemotherapy 6
Started | 3 (the patients received a total radiation dose of 57.2 Gy in this group) | 3 (the patients received a total radiation dose of 64.4 Gy in this group) | 3 (the patients received a total radiation dose of 71.6 Gy in this group) | 6 (the patients received a total radiation dose of 78.8 Gy in this group) | 13 (the patients received a total radiation dose of 86 Gy in this group) | 3 (the patients received a total radiation dose of 93.2 Gy in this group)
Completed | 3 (the patients received a total radiation dose of 57.2 Gy in this group) | 3 (the patients received a total radiation dose of 64.4 Gy in this group) | 3 (the patients received a total radiation dose of 71.6 Gy in this group) | 6 (the patients received a total radiation dose of 78.8 Gy in this group) | 13 (the patients received a total radiation dose of 86 Gy in this group) | 3 (the patients received a total radiation dose of 93.2 Gy in this group)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Radiochemotherapy 1: 3 Patients will be treated with radiation therapy 57.2 Gy.
  radiochemotherapy 1: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 7.2 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2, weekly; paclitaxel, 45-50 mg/m2, weekly
- Radiochemotherapy 2: 3 Patients will be treated with radiation therapy 64.4 Gy.
  radiochemotherapy 2: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 14.4 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Radiochemotherapy 3: 3 Patients will be treated with radiation therapy 71.6 Gy.
  radiochemotherapy 3: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 21.6 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Radiochemotherapy 4: 6 Patients will be treated with radiation therapy 78.8 Gy.
  radiochemotherapy 4: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 28.8 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Radiochemotherapy 5: 13 Patients will be treated with radiation therapy 86 Gy.
  radiochemotherapy 5: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 36 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
- Radiochemotherapy 6: 3 Patients will be treated with radiation therapy 93.2 Gy.
  radiochemotherapy 6: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 43.2 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Total: Total of all reporting groups
Arm/Group | Radiochemotherapy 1 | Radiochemotherapy 2 | Radiochemotherapy 3 | Radiochemotherapy 4 | Radiochemotherapy 5 | Radiochemotherapy 6 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 13 | 3 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 3 | 8 | 1 | 17
  >=65 years | 2 | 1 | 1 | 3 | 5 | 2 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 1 | 5 | 0 | 8
  Male | 2 | 3 | 2 | 5 | 8 | 3 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 3 | 3 | 3 | 6 | 13 | 3 | 31
Eastern Cooperative Oncology Group, ECOG performance status 0-1 [Count of Participants; unit: Participants] — GRADE ECOG PERFORMANCE STATUS
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants | 3 | 2 | 3 | 5 | 12 | 3 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) Occurring in Participants
Description: The DLTs were defined as grade >/=4 esophatitis, any other grade >/=3 nonhematological toxicity (except nausea and vomiting), or grade >/=4 hematological toxicity lasting more than 7 days, which are possibly, probably, or definitely associated with protocol treatment occurring during and after completion of the HFRT boost treatment.
Time Frame: 15 months
Measure: Number; unit: dose limiting toxicity
Groups:
- Arm 1: Radiochemotherapy 1: Patients will be treated with radiation therapy 57.2 Gy.
  radiochemotherapy 1: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 7.2 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
- Arm 2: Radiochemotherapy 2: Patients will be treated with radiation therapy 64.4 Gy.
  radiochemotherapy 2: concurrent radiochemotherapy: radiotherapy dose level 2: 50 Gy at 2 Gy/Fx/d, then 14.4 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
- Arm 3：Radiochemotherapy 3: Patients will be treated with radiation therapy 71.6 Gy.
  radiochemotherapy 3: concurrent radiochemotherapy: radiotherapy dose level 3: 50 Gy at 2 Gy/Fx/d, then 21.6 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
- Arm 4: Radiochemotherapy 4: Patients will be treated with radiation therapy 78.8 Gy.
  radiochemotherapy 4: concurrent radiochemotherapy: radiotherapy dose level 4: 50 Gy at 2 Gy/Fx/d, then 28.8 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
- Arm 5: Radiochemotherapy 5: Patients will be treated with radiation therapy 86 Gy.
  radiochemotherapy 5: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 36 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
- Arm 6: Radiochemotherapy 6: Patients will be treated with radiation therapy 93.2 Gy.
  radiochemotherapy 6: concurrent radiochemotherapy: radiotherapy dose level 6: 50 Gy at 2 Gy/Fx/d, then 43.2 Gy at 1.2 Gy/Fx/bid; concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly;
Arm/Group | Arm 1: Radiochemotherapy 1 | Arm 2: Radiochemotherapy 2 | Arm 3：Radiochemotherapy 3 | Arm 4: Radiochemotherapy 4 | Arm 5: Radiochemotherapy 5 | Arm 6: Radiochemotherapy 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 13 | 3
dose limiting toxicity | 0 | 0 | 0 | 1 | 0 | 2

2. Secondary Outcome: Local Failure
Description: Local failure will be assessed radiographically using endoscopy with biopsy, CT scan, and a positron emission computed tomography-CT scan. which was defined as persistence /recurrence of the tumor in the radiation therapy field.
Time Frame: 15 months
Population: the patients who completed the protocol treatment
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Radiochemotherapy 1: patients were be treated with radiation therapy 57.2 Gy
- Arm 2: Radiochemotherapy 2: patients were be treated with radiation therapy 64.4 Gy
- Arm 3: Radiochemotherapy 3: patients were be treated with radiation therapy 71.6 Gy
- Arm 4: Radiochemotherapy 4: patients were be treated with radiation therapy 78.8 Gy
- Arm 5: Radiochemotherapy 5: patients were be treated with radiation therapy 86 Gy
- Arm 6: Radiochemotherapy 6: patients were be treated with radiation therapy 93.2Gy
Arm/Group | Arm 1: Radiochemotherapy 1 | Arm 2: Radiochemotherapy 2 | Arm 3: Radiochemotherapy 3 | Arm 4: Radiochemotherapy 4 | Arm 5: Radiochemotherapy 5 | Arm 6: Radiochemotherapy 6
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 13 | 3
Participants | 0 | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 15 months
Groups:
- Arm 1: Radiochemotherapy 1: Patients will be treated with radiation therapy 57.2 Gy.
  radiochemotherapy 1: concurrent radiochemotherapy: radiotherapy dose level 1: 50 Gy at 2 Gy/Fx/d, then 57.2 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Arm 2: Radiochemotherapy 2: Patients will be treated with radiation therapy 64.4 Gy.
  radiochemotherapy 2: concurrent radiochemotherapy: radiotherapy dose level 2: 50 Gy at 2 Gy/Fx/d, then 14.4 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Arm 3: Radiochemotherapy 3: Patients will be treated with radiation therapy 71.6 Gy.
  radiochemotherapy 3: concurrent radiochemotherapy: radiotherapy dose level 3: 50 Gy at 2 Gy/Fx/d, then 21.6 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Arm 4: Radiochemotherapy 4: Patients will be treated with radiation therapy 78.8Gy.
  radiochemotherapy 4: concurrent radiochemotherapy: radiotherapy dose level 4: 50 Gy at 2 Gy/Fx/d, then 28.8 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Arm 5: Radiochemotherapy: Patients will be treated with radiation therapy 36 Gy.
  radiochemotherapy 5: concurrent radiochemotherapy: radiotherapy dose level 5: 50 Gy at 2 Gy/Fx/d, then 36 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
- Arm 6: Radiochemotherapy 6: Patients will be treated with radiation therapy 93.2 Gy.
  radiochemotherapy 6: concurrent radiochemotherapy: radiotherapy dose level 6: 50 Gy at 2 Gy/Fx/d, then 43.2 Gy at 1.2 Gy/Fx/bid concurrent chemotherapy: carboplatin, area under the curve (AUC) 1.5-2,weekly; paclitaxel, 45-50 mg/m2, weekly
Arm/Group | Arm 1: Radiochemotherapy 1 | Arm 2: Radiochemotherapy 2 | Arm 3: Radiochemotherapy 3 | Arm 4: Radiochemotherapy 4 | Arm 5: Radiochemotherapy | Arm 6: Radiochemotherapy 6
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/13 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/13 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/6 | 11/13 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Radiochemotherapy 1 (N=3) | Arm 2: Radiochemotherapy 2 (N=3) | Arm 3: Radiochemotherapy 3 (N=3) | Arm 4: Radiochemotherapy 4 (N=6) | Arm 5: Radiochemotherapy (N=13) | Arm 6: Radiochemotherapy 6 (N=3)
grade 3 pneumotitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
grade 5 esophageal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Radiochemotherapy 1 (N=3) | Arm 2: Radiochemotherapy 2 (N=3) | Arm 3: Radiochemotherapy 3 (N=3) | Arm 4: Radiochemotherapy 4 (N=6) | Arm 5: Radiochemotherapy (N=13) | Arm 6: Radiochemotherapy 6 (N=3)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 3 (3) | 5 (5) | 11 (11) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03082586/Prot_SAP_ICF_000.pdf